CLINICAL TRIAL: NCT01301508
Title: A Multi-Center, Randomized, Double-Blind, Vehicle-Controlled, Bilateral Study of the Safety and Efficacy of Topically Applied AN2898 and AN2728 in the Treatment of Patients With Mild-to-Moderate Atopic Dermatitis
Brief Title: Efficacy and Safety of AN2898 and AN2728 Topical Ointments to Treat Mild-to-Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN2898-AD-202; C3471001 (Other: Pfizer)
Record Dates: First submitted 2011-02-17; First posted 2011-02-23 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AN2898 ointment, 1%, vs. ointment vehicle (Experimental): AN2898 ointment applied twice daily for 6 weeks to one target lesion, and AN2898 ointment vehicle applied twice daily for 6 weeks to a second target lesion.
  Treatments will be randomly assigned to target lesions A and B.
  Interventions: Drug: AN2898 ointment, 1%; Drug: AN2898 ointment vehicle
- AN2728 ointment, 2%, vs. ointment vehicle (Experimental): AN2728 ointment applied twice daily for 6 weeks to one target lesion, and AN2728 ointment vehicle applied twice daily for 6 weeks to a second target lesion.
  Treatments will be randomly assigned to target lesions A and B.
  Interventions: Drug: AN2728 ointment, 2%; Drug: AN2728 ointment vehicle

INTERVENTIONS:
Drug: AN2728 ointment, 2% — AN2728 ointment, 2%, applied twice daily for 6 weeks
  Arms: AN2728 ointment, 2%, vs. ointment vehicle
Drug: AN2898 ointment, 1% — AN2898 ointment, 1%, applied twice daily for 6 weeks
  Arms: AN2898 ointment, 1%, vs. ointment vehicle
Drug: AN2898 ointment vehicle — AN2898 ointment vehicle applied twice daily for 6 weeks
  Arms: AN2898 ointment, 1%, vs. ointment vehicle
Drug: AN2728 ointment vehicle — AN2728 ointment vehicle applied twice daily for 6 weeks
  Arms: AN2728 ointment, 2%, vs. ointment vehicle

SUMMARY:
The purpose of this study is to determine whether AN2898 and AN2728 ointments are safe and effective treatments for mild-to-moderate atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of atopic dermatitis that has been clinically stable for ≥1 month
* Total body surface area (BSA) of atopic dermatitis involvement ≤35%, excluding involvement of the face, scalp, and groin
* Presence of two (2) comparable target lesions
* Willing and able to apply study medications as directed, comply with study instructions, and commit to attending all visits
* Females of childbearing potential must use at least one highly effective method of birth control. Males with partners of childbearing potential should inform them of their participation in this clinical study and use highly effective methods of birth control during the study.

Exclusion Criteria:

* Concurrent or recent use of certain topical or systemic medications or phototherapy without a sufficient washout period
* Active or potentially recurrent dermatologic condition other than atopic dermatitis in the target lesion area that may confound evaluation
* Significant confounding conditions as assessed by study doctor
* History or evidence of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis)
* Participated in any other trial of an investigational drug or device within 30 days or participation in a research study concurrent with this study
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11-11 (Actual); Study Completion 2011-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- Australia (13):
  - Anacor Investigational Site, Kogarah, New South Wales
  - Anacor Investigational Site, Brisbane, Queensland
  - Anacor Investigational Site, Woolloongabba, Queensland
  - Anacor Investigational Site, Adelaide, South Australia
  - Anacor Investigational Site, Box Hill, Victoria
  - Anacor Investigational Site, Carlton, Victoria
  - Anacor Investigational Site, Clayton, Victoria
  - Anacor Investigational Site, Fitzroy, Victoria
  - Anacor Investigational Site, Parkville, Victoria
  - Anacor Investigational Site, Fremantle, Western Australia
  - Anacor Investigational Site, Nedlands, Western Australia
  - Anacor Investigational Site, Subiaco, Western Australia
  - Anacor Investigational Site, Victoria Park, Western Australia

REFERENCES:
- [Derived] Murrell DF, Gebauer K, Spelman L, Zane LT. Crisaborole Topical Ointment, 2% in Adults With Atopic Dermatitis: A Phase 2a, Vehicle-Controlled, Proof-of-Concept Study. J Drugs Dermatol. 2015 Oct;14(10):1108-12. PMID 26461821

RESULTS

PARTICIPANT FLOW:
Groups:
- AN2898 Ointment, 1% + Ointment Vehicle: Participants with mild to moderate atopic dermatitis (AD) applied AN2898 ointment, 1 percent (%) to one target lesion (active lesion), topically twice daily from Day 1 to 42 and AN2898 ointment vehicle applied twice daily from Day 1 to 42 to a second target lesion (vehicle lesion). Target lesions were identified at Baseline (Day 1) by investigator.
- AN2728 Ointment, 2% + Ointment Vehicle: Participants with mild to moderate AD applied AN2728 ointment, 2% to one target lesion (active lesion), topically twice daily from Day 1 to 42 and AN2728 ointment vehicle applied twice daily from Day 1 to 42 to a second target lesion (vehicle lesion). Target lesions were identified at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Started | 21 | 25
Completed | 20 | 22
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all randomized participants with confirmed usage of the study medication.
Groups:
- AN2898 Ointment, 1% + Ointment Vehicle: Participants with mild to moderate AD applied AN2898 ointment, 1% to one target lesion (active lesion), topically twice daily from Day 1 to 42 and AN2898 ointment vehicle applied twice daily from Day 1 to 42 to a second target lesion (vehicle lesion). Target lesions were identified at Baseline (Day 1) by investigator.
- Total: Total of all reporting groups
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle | Total
Number analyzed (Participants) | 21 | 25 | 46
Age, Customized [Count of Participants; unit: Participants]
  18 to 65 years | 21 | 22 | 43
  Greater Than 65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 10 | 15 | 25

OUTCOME MEASURES:

1. Primary Outcome: Atopic Dermatitis Severity Index (ADSI) Score at Baseline (Day 1)
Description: ADSI score was used to measure the severity of participant's atopic dermatitis (AD) affected lesion. It evaluated 5 signs of AD (erythema, pruritus, exudation, excoriation and lichenification) in each lesion. Each sign was rated by investigator on a scale of 0 (none) to 3 (severe), where higher score indicated more severe condition. Total ADSI score for each lesion was sum of scores of the 5 signs and ranged from 0 (none) to 15 (most severe), where higher score indicated more severe condition.
Time Frame: Baseline (Day 1)
Population: The intent-to-treat (ITT) population included all randomized participants who received study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Number analyzed (Participants) | 21 | 25
units on a scale
  Active Lesion | 8.0 (1.21) | 8.3 (1.77)
  Vehicle Lesion | 8.0 (1.24) | 8.4 (1.75)

2. Primary Outcome: Atopic Dermatitis Severity Index (ADSI) Score at Day 14
Description: ADSI score was used to measure the severity of participant's AD affected lesion. It evaluated 5 signs of AD (erythema, pruritus, exudation, excoriation and lichenification) in each lesion. Each sign was rated by investigator on a scale of 0 (none) to 3 (severe), where higher score indicated more severe condition. Total ADSI score for each lesion was sum of scores of the 5 signs and ranged from 0 (none) to 15 (most severe), where higher score indicated more severe condition.
Time Frame: Day 14
Population: ITT population included all randomized participants who received study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Number analyzed (Participants) | 21 | 25
units on a scale
  Active Lesion | 3.8 (1.98) | 4.0 (2.54)
  Vehicle Lesion | 5.4 (2.73) | 5.6 (3.17)

3. Primary Outcome: Atopic Dermatitis Severity Index (ADSI) Score at Day 28
Description: as for outcome 2
Time Frame: Day 28
Population: ITT population included all randomized participants who received study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Number analyzed (Participants) | 21 | 25
units on a scale
  Active Lesion | 2.6 (1.78) | 2.8 (2.30)
  Vehicle Lesion | 4.3 (3.54) | 5.1 (3.33)

4. Primary Outcome: Atopic Dermatitis Severity Index (ADSI) Score at Day 42
Description: as for outcome 2
Time Frame: Day 42
Population: ITT population included all randomized participants who received study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Number analyzed (Participants) | 21 | 25
units on a scale
  Active Lesion | 3.5 (3.75) | 3.0 (2.98)
  Vehicle Lesion | 3.1 (3.12) | 4.6 (3.57)

5. Primary Outcome: Percentage of Participants With Decrease From Baseline in Atopic Dermatitis Severity Index (ADSI) Score at Day 28
Description: ADSI score was used to measure the severity of participant's AD affected lesion. It evaluated 5 signs of AD (erythema, pruritus, exudation, excoriation and lichenification) in each lesion. Each sign was rated by investigator on a scale of 0 (none) to 3 (severe), where higher score indicated more severe condition. Total ADSI score for each lesion was sum of scores of the 5 signs and ranged from 0 (none) to 15 (most severe), where higher score indicated more severe condition. Percentage of participants in whom the active lesion (ointment treated) achieved a greater decrease from baseline to Day 28 in ADSI as compared to vehicle lesion (vehicle treated) and, in whom the vehicle lesion (vehicle treated) achieved a greater decrease from baseline to Day 28 as compared to active lesion (ointment treated) were reported in this outcome measure.
Time Frame: Baseline (Day 1), Day 28
Population: ITT population included all randomized participants who received study medication.
Measure: Number; unit: percentage of participants
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Number analyzed (Participants) | 21 | 25
percentage of participants
  Greater Decrease in Active Lesion | 71.4 | 68.0
  Greater Decrease in Vehicle Lesion | 14.3 | 20.0
Statistical Analysis 1: Comparison: AN2898 Ointment, 1% + Ointment Vehicle; Test type: Superiority or Other; p = 0.008, Two-sided sign test — p-value was calculated for the statistical significant difference between greater decrease in vehicle lesion and greater decrease in active lesion for the AN2898 Topical Ointment, 1% + Ointment Vehicle group
Statistical Analysis 2: Comparison: AN2728 Ointment, 2% + Ointment Vehicle; Test type: Superiority or Other; p = 0.017, Two-sided sign test — p-value was calculated for the statistical significant difference between greater decrease in vehicle lesion and greater decrease in active lesion for the AN2728 Topical Ointment, 2% + Ointment Vehicle group

6. Other Pre Specified Outcome: Percentage of Participants With Decrease From Baseline in Atopic Dermatitis Severity Index (ADSI) Score at Day 14 and 42
Description: ADSI score was used to measure the severity of participant's AD affected lesion. It evaluated 5 signs of AD (erythema, pruritus, exudation, excoriation and lichenification) in each lesion. Each sign was rated by investigator on a scale of 0 (none) to 3 (severe), where higher score indicated more severe condition. Total ADSI score for each lesion was sum of scores of the 5 signs and ranged from 0 (none) to 15 (most severe), where higher score indicated more severe condition. Percentage of participants in whom the active lesion (ointment treated) achieved a greater decrease from baseline to Days 14, 42 in ADSI as compared to vehicle lesion (vehicle treated) and, in whom the vehicle lesion (vehicle treated) achieved a greater decrease from baseline to Days 14, 42 as compared to active lesion (ointment treated) were reported in this outcome measure.
Time Frame: Baseline (Day 1), Day 14, Day 42
Population: ITT population included all randomized participants who received study medication.
Measure: Number; unit: percentage of participants
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Number analyzed (Participants) | 21 | 25
percentage of participants
  Greater Decrease in Active Lesion: Day 14 | 57.1 | 64.0
  Greater Decrease in Vehicle Lesion: Day 14 | 14.3 | 20.0
  Greater Decrease in Active Lesion: Day 42 | 47.6 | 64.0
  Greater Decrease in Vehicle Lesion: Day 42 | 42.9 | 20.0

7. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. The SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death, initial or prolonged inpatient hospitalization, life-threatening experience (immediate risk of dying), persistent or significant disability or incapacity, congenital anomaly. Treatment-emergent were events between first dose of study medication and up to the end of study treatment (Day 42) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious adverse events.
Time Frame: Baseline (Day 1) up to Day 42
Population: Safety analysis population included all randomized participants with confirmed usage of the study medication.
Measure: Number; unit: participants
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Number analyzed (Participants) | 21 | 25
participants
  AEs | 11 | 11
  SAEs | 0 | 0

ADVERSE EVENTS:
Arm/Group | AN2898 Ointment, 1% + Ointment Vehicle | AN2728 Ointment, 2% + Ointment Vehicle
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/25
Other Adverse Events (participants affected / at risk) | 11/21 | 11/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AN2898 Ointment, 1% + Ointment Vehicle (N=21) | AN2728 Ointment, 2% + Ointment Vehicle (N=25)
Ear pain (Ear and labyrinth disorders) | 0 | 1
Application site erythema (General disorders) | 1 | 1
Application site irritation (General disorders) | 0 | 1
Application site pain (General disorders) | 0 | 1
Application site pruritus (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Application site cellulitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 6
Urinary tract infection (Infections and infestations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 1 | 2
Migraine (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.